CLINICAL TRIAL: NCT06477484
Title: Blood-based Biomarkers for Early Alzheimer's Disease Screening
Brief Title: Blood Biomarkers for Screening of Alzheimer's Disease
Status: Recruiting | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2024SF35
Record Dates: First submitted 2024-06-06; First posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Alzheimer's Disease; Blood Biomarkers
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- different stages of individuals with Alzheimer's disease
  Interventions: Diagnostic Test: Blood biomarker

INTERVENTIONS:
Diagnostic Test: Blood biomarker — Blood biomarker

SUMMARY:
The goal of this observational study is to estimate the screen performance of blood biomarkers of interest (Aβ40 and Aβ42, P-Tau181, P-Tau217, GFAP and NfL) in patients with Alzheimer's disease (AD), mild cognitive impairment due to AD, and cognitively normal individuals. The main questions it aims to answer are:

* to identify core blood biomarker suitable for early screening of AD.
* to establish a comprehensive model for the early identification of AD.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years;
* AD (meets the 2011 NIA-AA AD diagnostic criteria), or MCI (meets the 2004 Peterson MCI diagnostic criteria), or cognitively normal subjects;
* Signed informed consent form.

Exclusion Criteria:

* The presence of other disorders that can cause cognitive impairment;
* Unable to cooperate with the completion of cognitive assessment;
* Refusal to draw blood.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Alzheimer's disease, mild cognitive impairment due to AD, and cognitively normal individuals.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2024-06-18 (Actual); Primary Completion 2026-03-26 (Estimated); Study Completion 2026-03-26 (Estimated)

PRIMARY OUTCOMES:
Evaluate the diagnostic accuracy of blood biomarkers of Aβ42, Aβ40, Aβ42/Aβ40, P-Tau181, P-Tau217, GFAP and NfL. | 2 years

SECONDARY OUTCOMES:
Evaluate the diagnostic accuracy of a comprehensive model combined with core blood biomarkers and clinical information. | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China